CLINICAL TRIAL: NCT01374594
Title: Importance of Meal Fat Content and Gall Bladder Emptying for Postprandial GLP-1 Secretion in Type 2 Diabetes Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, David P. Sonne, MD, University Hospital, Gentofte, Copenhagen
Other Study IDs: GAL-INK II
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Biospecimen Retention: blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy adults
- Type 2 diabetes

SUMMARY:
PURPOSE

The goal of the present project is to unravel the importance of bile acid-induced GLP-1 secretion (via the G protein-coupled receptor TGR5) in human physiology.

In the present study the investigators examine the GLP-1 secretion in healthy subjects and in Type 2 Diabetes Mellitus (T2DM) patients. The investigators hypothesize that patients with T2DM of relatively long duration will be characterized by reduced gall bladder emptying, and, consequently, reduced intestinal TGR5 activation; resulting in attenuated postprandial GLP-1 responses (primary endpoint).

ELIGIBILITY:
Inclusion Criteria: (Healthy)

* HbA1 < 6 %
* Normal haemoglobin levels
* Informed content

Inclusion Criteria: (T2DM)

* T2DM > 5 years
* Normal haemoglobin levels
* Informed content

Exclusion Criteria: (T2DM)

* Treatment with insulin, DPP-IV inhibitor or GLP-1 analogues
* Obesity (BMI > 30)
* Age > 70 years
* Gastrointestinal disease
* Nephropathy
* Liver disease
* Medication which cannot be on hold for 12h
* Gastrointestinal surgery

Exclusion Criteria: (Healthy)

* 1st degree relatives with diabetes
* Obesity (BMI > 30)
* Age > 70 years
* Gastrointestinal disease
* Nephropathy
* Liver disease
* Medication which cannot be on hold for 12h
* Gastrointestinal surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects and type 2 diabetes patients (T2DM)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
GLP-1 secretion | Postprandial

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte University Hospital, Hellerup, Denmark

REFERENCES:
- [Derived] Sonne DP, van Nierop FS, Kulik W, Soeters MR, Vilsboll T, Knop FK. Postprandial Plasma Concentrations of Individual Bile Acids and FGF-19 in Patients With Type 2 Diabetes. J Clin Endocrinol Metab. 2016 Aug;101(8):3002-9. doi: 10.1210/jc.2016-1607. Epub 2016 Jun 7. PMID 27270475
- [Derived] Sonne DP, Vilsboll T, Knop FK. Pancreatic Amylase and Lipase Plasma Concentrations Are Unaffected by Increments in Endogenous GLP-1 Levels Following Liquid Meal Tests. Diabetes Care. 2015 May;38(5):e71-2. doi: 10.2337/dc14-2751. No abstract available. PMID 25908158